CLINICAL TRIAL: NCT04711876
Title: Study of the Inflammatory Response to Enterovirus Meningitis in Newborns, Infants and Children, as Assessed by Cytokine Levels in Blood and Cerebrospinal Fluid. Case-control Comparison Using an Existing Cohort.
Brief Title: Characterization of Cytokines Expression During Enterovirus Meningitis in Paediatric Populations.
Acronym: Bledi-Cytokine
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Laboratory of virology, National Enterovirus and parechovirus Reference Center, University Hospital of Clermont-Ferrand (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020 ARCHIMBAUD Bledi-Cytokine
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Meningitis Enterovirus
Keywords: Enterovirus infection; Cytokine expression; Paediatric population; Blood; Cerebrospinal fluid; Inflammatory; Meningitis viral
MeSH Terms: conditions — Enterovirus Infections; Meningitis, Viral | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood and CSF taken from paediatric patient during hospitalisation for suspicion of meningitis (Sample taken from 2015 and 2016 according to the BLEDI Study)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test group with enterovirus meningitis: Level of Cytokine in blood and CSF for Patient with RT-PCR-EV +
  Interventions: Biological: Cytokine level in blood and CSF
- Control group with no enterovirus meningitis: Level of Cytokine in blood and CSF for Patient with RT-PCR-EV -
  Interventions: Biological: Cytokine level in blood and CSF

INTERVENTIONS:
Biological: Cytokine level in blood and CSF — Measure of cytokine level

SUMMARY:
Enteroviruses (EV) are the most frequent cause of acute meningitis in the paediatric population. Detection of enterovirus in cerebrospinal fluid (CSF) specimens by Polymerase Chain Reaction (PCR) is the gold standard diagnostic test. Recently, our laboratory published the BLEDI study which highlighted the interest of detecting EV in the blood of the paediatric population : (i) EV was found in more than a quarter of cases in the blood of infants admitted to hospital with isolated fever and (ii) detection of EV was more frequent in the blood than in CSF in neonates and infants with isolated fever, sepsis or meningitis. However, the pathophysiology of EV infections is poorly understood and little work has been done on the inflammatory response to these infections. In EV meningitis, the inflammatory response has been studied primarily in children infected with enterovirus A71 (EV-A71). Indeed, in these children, inappropriate cytokine secretion (cytokine storm) leads to severe neurological and cardiopulmonary damage, which can progress to death. The study of the inflammatory response during meningitis due to other types of EV remains poorly

The objective of BLEDI-CYTOKINES (ancillary study of the BLEDI study) is to study the inflammatory response during EV meningitis in neonates, infants and children, as assessed by cytokine levels in blood and cerebrospinal fluid, by comparing case-controls from an existing cohort.

DETAILED DESCRIPTION:
EVs are characterized by their high genetic variability, with more than 120 types described to date. They are involved in mild infections, such as febrile syndromes that may be associated with respiratory and cutaneous manifestations. However, these viruses are also involved in more severe infections of the nervous system. In children infected with EV-A71, which causes mild epidemics of foot-and-mouth disease, inappropriate cytokine secretion (cytokine storm) leads to severe neurological and cardiopulmonary complications that can progress to death in children (<5 years of age) in Asia. Many studies have focused on the inflammatory response to EV-A71 infections: some cytokines (Tumor Necrose Factor (TNF), INterFeron (INF), InterLeukine (IL)1, IL6, IL10, eotaxin,...) dosed in CSF have been associated with severe EV-A71 infections (2,5,6). Recently, a Japanese study showed an overexpression of IL-6 in the blood of children with EV-A71 foot-hand-mouth syndrome. The authors defined that a level of IL-6 ≥ 66 pg/mL could be a prognostic marker of progression to aseptic meningitis (6). In EV (other than EV-A71) meningitis, pro-inflammatory cytokines such as IL6, IL8, and INF are produced in the acute phase in CSF to control the infection, and then they decline and anti-inflammatory cytokines such as IL10 are synthesized (7). In addition, studies have shown that the production of some cytokines is greater in severe EV infections: for example, the production of IL4 and IL5 is greater in EV encephalitis than in EV skin infections (8).

However, there are very few comparative studies of cytokine expression in blood and CSF. In addition, little work has been done to study cytokine expression in meningitis due to EV other than EV-A71. In young children, these meningitis may also be complicated by encephalitis, myelitis, and even flaccid paralysis (including poliomyelitis) (2-4). The pathophysiology of these severe EV infections is currently unknown. In addition, no preventive vaccine is available against these infections (other than polio vaccine), nor are there effective curative antivirals for severe EV infections.

ELIGIBILITY:
Inclusion Criteria:

* Patients with proven enterovirus meningitis (RT- PCR EV positive)
* Control patients admitted for suspected meningitis infection but for whom the bacteriological (LCS culture/ blood culture negative) and virological diagnosis (testing for enteroviruses (RT-PCR negative) and parechoviruses (viruses responsible for symptoms similar to those of EVs) is negative

Exclusion Criteria:

For patients with EV meningitis, we will exclude:

* patients with co-infection
* haemorrhagic CSF samples
* samples (CSF or blood) for which we do not have access to EV viral load results
* samples (CSF or blood) for which we do not have access to the EV genotyping results

For patients in the control group (without EV meningitis), we will exclude :

* Samples from patients with an infection (viral or bacterial) in the control group.
* haemorrhagic CSF samples
* CSF samples with pleocytosis (presence of CSF leucocytes).
* Blood samples with high CRP (CRP>15mg/L).

Ages: 1 Day to 16 Years | Sex: All
Age Groups: Child
Study Population: Paediatric patient with suspicion of meningitis
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Expression of cytokine in blood | Day 1
  Level of cytokine in blood
Expression of cytokine in cerebrospinal fluid | Day 1
  Level of cytokine in cerebrospinal fluid

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Clermont Ferrand, Clermont-Ferrand, AURA, France

REFERENCES:
- [Background] Lafolie J, Labbe A, L'Honneur AS, Madhi F, Pereira B, Decobert M, Adam MN, Gouraud F, Faibis F, Arditty F, Marque-Juillet S, Guitteny MA, Lagathu G, Verdan M, Rozenberg F, Mirand A, Peigue-Lafeuille H, Henquell C, Bailly JL, Archimbaud C; Blood Enterovirus Diagnosis Infection (BLEDI) in paediatric population study team. Assessment of blood enterovirus PCR testing in paediatric populations with fever without source, sepsis-like disease, or suspected meningitis: a prospective, multicentre, observational cohort study. Lancet Infect Dis. 2018 Dec;18(12):1385-1396. doi: 10.1016/S1473-3099(18)30479-1. Epub 2018 Oct 30. PMID 30389482